CLINICAL TRIAL: NCT00083356
Title: Bradykinin-1 Receptor and Kinin Induction in a Clinical Model of Tissue Injury
Brief Title: Bradykinin Receptors and Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040182; 04-NR-0182
Record Dates: First submitted 2004-05-21; First posted 2004-05-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-02

CONDITIONS: Tooth, Impacted
Keywords: Pain; Kinins; Inflammation; Gene Expression; Oral Surgey; Bradykinin B1 Receptors; Acute Peripheral Inflammation; Inflammatory Gene Expression; Wisdom Teeth; Third Molar Extraction
MeSH Terms: conditions — Tooth, Impacted; Pain; Inflammation

INTERVENTIONS:
Procedure: Wisdom tooth extraction

SUMMARY:
This study will examine whether bradykinin receptors are produced at the site of wisdom tooth extraction and if they contribute to the amount of inflammation and pain that follows surgery. Bradykinin is a molecule produced by enzymes at the site of an injury and then binds to receptors to cause pain. The study will also evaluate the role of genetic factors in the production of bradykinin and their receptors and the pain associated with minor surgical procedures.

Patients between 16 and 35 years of age who are referred to the NIH dental clinic for removal of two wisdom teeth may be eligible for this study. Candidates must be in good health and must not be allergic to aspirin, non-steroidal anti-inflammatory drugs, sulfites, or amide anesthetics. They will be screened with a medical history and oral examination, including x-rays to confirm the need for wisdom tooth extraction.

On the morning of surgery following an overnight fast, participants have a blood sample drawn to extract DNA for gene studies. Just before surgery, they are given an intravenous (IV) sedative to induce drowsiness and a local anesthetic to numb the mouth. They are also given IV either Ketorolac, a non-steroidal anti-inflammatory drug, or placebo, a look-alike medication with no active ingredient. After the extractions, a small piece of plastic tubing is placed in both extraction sites, and every 20 minutes for the next 3 hours inflammatory fluid is collected from the tubing for measuring chemicals believed to cause pain and swelling. Patients rate their pain by answering pain-related questions every 20 minutes. Patients who have pain that is not relieved by the study medication (Ketorolac or placebo) are given, upon request, 50 mg of the pain reliever tramadol (Ultram). Patients remain in the clinic for at least 3 hours and no more than 7 hours after surgery in order for monitoring the effects of the study drugs as the local anesthetic wears off.

Patients undergo two biopsies during the study - one before and one after the extraction - to measure any changes in chemicals produced in response to the surgery. The second biopsy is done either 3, 7, or 24 hours after the extraction. Patients in the 3- and 7-hour groups are given a small dose of local anesthetic in the gum for the second biopsy and remain in the clinic until the biopsy is done; those in the 24-hour group are given forms to record pain ratings at home and return to the clinic the following morning for a 2-hour follow-up visit. All patients are given standard pain medication (flurbiprofen) to take at home.

DETAILED DESCRIPTION:
Bradykinin B1 receptors and their natural agonists are known to be rapidly induced in local tissues by a variety of inflammatory stimuli. Preclinical evidence, demonstrating that interruption of B1 receptor function causes analgesia under a variety of conditions, has been well established using selective antagonists and genetically modified mice. Accordingly, efforts are underway in several laboratories to develop novel B1 receptor antagonists as potential novel analgesic agents. The proposed studies will examine the kinetics of local induction of B1 receptors and kinin formation in a common situation of acute inflammatory pain in humans - tooth extraction. In addition, an examination of expression of additional genes of interest under these conditions using microarray analysis will be conducted.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female volunteers referred for third molar extraction willing to undergo 2 or 3 visits: 1 screening visit; 1 surgical appointment; and a possible follow-up research-related appointment

Between the ages of 16 to 35 years (based upon eruption patterns and age-related complications associated with surgical extraction of third molars

In general good health- American Society of Anesthesiologists (ASA) status I or II (healthy subjects based upon criteria for safe administration of out-patient conscious sedation)

Willing to undergo observation period for three hours postoperatively

Ability to complete a 100 mm visual analog scale and a category scale every 20 minutes for the first 3 postoperative hours

Willing to have a microdialysis probe placed beneath the surgical flap during the first 3 hours post-surgery

Willing to have a preoperative biopsy on the day of surgery, and a postoperative biopsy either at 3, 7 or 24 hours following surgery

Willing to return, if needed, 24 hours post-operation for the postoperative biopsy

Must have two lower partial (rating is equal to 3) or fully impacted (rating is equal to 4) wisdom teeth (mandibular third molars)

As assessed at the screening visit, the sum of the mandibular third molar surgical difficulty ratings must be between 6 to 8 in order to evaluate subjects experiencing similar pain levels

EXCLUSION CRITERIA:

Patients who are allergic to aspirin, NSAIDs, sulfites, or amide anesthetics

Patients who have had asthma, or hives

Patients who are pregnant or nursing

Patients with history of peptic ulcers and/or GI bleeding

Chronic use of medications confounding the assessment of the inflammatory response or analgesia, for example, NSAIDs, COX-2 inhibitors, antihistamines, steroids, antidepressants

Patients who have clinical signs suggestive of infection, inflammation, or pre-existing pain at either extraction site

Patients with severe kidney disease

Patients who are taking any of the following drugs: ACE inhibitor; potassium sparing diuretics; aspirin on a near daily basis; coumadin or other blood thinners

Patients who are taking drugs known to inhibit P450 2C9 and drugs metabolized by P450 2D6

Unusual surgical difficulty (determined from panoramic radiograph or during the actual surgery)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2004-05; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Nursing Research (NINR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Walker K, Perkins M, Dray A. Kinins and kinin receptors in the nervous system. Neurochem Int. 1995 Jan;26(1):1-16; discussion 17-26. doi: 10.1016/0197-0186(94)00114-a. PMID 7787759
- [Background] Ahluwalia A, Perretti M. B1 receptors as a new inflammatory target. Could this B the 1? Trends Pharmacol Sci. 1999 Mar;20(3):100-4. doi: 10.1016/s0165-6147(99)01321-8. PMID 10203864
- [Background] Bock MG, Longmore J. Bradykinin antagonists: new opportunities. Curr Opin Chem Biol. 2000 Aug;4(4):401-6. doi: 10.1016/s1367-5931(00)00107-1. PMID 10959767